CLINICAL TRIAL: NCT04429763
Title: Safety and Efficacy of Mesenchymal Stem Cells in the Management of Severe COVID-19
Brief Title: Safety and Efficacy of Mesenchymal Stem Cells in the Management of Severe COVID-19 Pneumonia
Acronym: CELMA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Trustem (Industry)
Collaborators: Fundación Universitaria de Ciencias de la Salud (Other); Hospital de San Jose (Other); Hospital Infantil Universitario de San Jose (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202001
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: Mesenchymal Stem Cells; Umbilical Cord
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: It will be included 30 patients, randomly assigned by centralized electronic sequence of assignation, for the application of a single dosis of 1*10^6 cells/Kg or placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Usual tratment for COVID-19 plus MSC
  Interventions: Biological: Umbilical cord derived mesenchymal stem cells
- Control (Placebo Comparator): Usual treatment for COVID-19
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Umbilical cord derived mesenchymal stem cells — One dosis of 1*10^6 cells/Kg
  Arms: Experimental
Biological: Placebo — Placebo
  Arms: Control

SUMMARY:
The disease caused by the new coronavirus, SARS-CoV-2, called COVID-19, it has considered a worldwide pandemia by the WHO. Suddently, it produces a lot of patients severe ill, in a little geographic area, that could surpase the resourses of the any health system in the world.

There is no documentation of an effective alternative for the treatment of the severe ill patients, that can reduce the mortality or the adverse events suffered by these people.

It is has suggested the usefulness of the Mesenchymal Stem cells (MSC) for the management of these patients, thanks to their direct and indirect antiviral capacity, and its potency as immunomodulator, that could ameliorate the lung disease and the severity of COVID-19.

DETAILED DESCRIPTION:
Objetive:

Evaluate the effect of MSC derived from human umbilical cord compared with placebo, over the clinical progresion and mortality of hospitalized COVID-19 patients.

Metodology:

Fase II, controled clinical trial, double blinded, compared with placebo, with paralel groups, and one to one asignation. It will be included patients between 18 and 79 years old, hositalized in general room (respiratory isolation area) with confirmed COVID-19 diagnosis. It will be excluded those who have indication for management in Intensive Care Unit, have any condition that seriusly affect their survival, pregnant whomen or breast feeding, those who have an advanced hearth failure, HIV infected, those who have a bacterial or fungal uncontroled infection, those who require permanent immunosupresive therapy or have had an organ trasplant, those who have no possibility to sign the informed consent format or are involved in another clinical trial with drugs or interventions.

It will vinculate 30 patients randomly assigned, by centralized electronic assignation sequence, for the experimental group who will received 1*10^6 cells/Kg extracted from human umbilical cord or to placebo group.

The primary result it will be a composed point of time to the occurrence of the clinical detriment or the death (the first that occurs) and the secondary result will be the components of each primary point, the clinical recovery, the time to the time to the discharge from the hospital, and the clinical follow-up, including respiratory function, and markers of inflammation, haematological and kidney, in addition of the safety markers.

It will be done a comparison of the incidence rates, by ratio of incidence rates and their respective confidence interval. It will be construct Kaplan-Meier curves that will compared by the statics of logaritmic rank (log-rank test).

It will be developed a multivariate analysis, with the Cox proportional risks methodology, estimating the Hazard Ratio epidemiologic.

ELIGIBILITY:
Inclusion Criteria:

* Severe COVID-19.
* Infection confirmed by PCR test.
* Hospitalized in general room (respiratory isolation area).

Exclusion Criteria:

* Shock or multiorgan disfunction that require continous vital signs monitorization
* Punctuation equal or more than 7 in the National Early Warning Score (NEWS) - 2 scale.
* Condition that seriously affects the patient survival expectancies, including any active cancer, hemorragia, any blood disease or severe malnutrition.
* Pregnant women or breast feeding.
* Advanced hearth failure.
* VIH/AIDS.
* Bacterial or fungical uncontroled infection.
* Permanente use of immunosupresants or have had received an organ trasnplanted in the past six months.
* Imposibility to sign the informent consent format.
* Patients involved in another clinical trial with drugs or interventions.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Clinical deterioration or death | 4 weeks
  Change in two or more degrees in the NEWS scale

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Sánchez-Vanegas, MD, PhD, Study Chair — Fundación Universitaria de Ciencias de la Salud; Carlos Escobar-Soto, MD, PhD, Study Director — Trustem

IPD SHARING:
Plan to Share IPD: No